CLINICAL TRIAL: NCT06297967
Title: Acetic Acid in Cutaneous Ulcers. A Randomized Controlled Trial
Brief Title: Acetic Acid 2% Solution for Skin Ulcers
Acronym: ECA-AA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSAPG-33
Record Dates: First submitted 2024-02-23; First posted 2024-03-07 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Ulcer, Skin
Keywords: Skin Ulcer; Acetic Acid; Biofilms
MeSH Terms: conditions — Skin Ulcer | interventions — Acetic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetic Acid (Experimental): Topic application of a Acetic Acid 2% solution for 15 min, typically administered every 24h. The frequency of the treatments may be modified according to the evolution of the lesion at the discretion of the nurse in charge of the treatments
  Interventions: Drug: Acetic Acid
- Control group (Active Comparator): Topic application of Prontosan® for 15 min, typically administered every 24h. The frequency of the treatments may be modified according to the evolution of the lesion at the discretion of the nurse in charge of the treatments
  Interventions: Drug: Prontosan

INTERVENTIONS:
Drug: Acetic Acid — The intervention treatment will consist of cleaning with water and soap, application of a compress soaked in 2% dilution of glacial acetic acid (CAS 64-19-7) for 15 minutes, irrigation with distilled water, application of peri-ulcer barrier cream or spray, and the application of ActicoatⓇ on the ulcer bed. Depending on the amount of exudate, more or less alginate will be added as a secondary dressing. A tertiary dressing of polyurethane foam or bandage will be applied according to the area and the nurse's discretion.
  Other Names: Acetic Acid 2%
  Arms: Acetic Acid
Drug: Prontosan — The treatment includes ulcer cleansing with water and soap, application of ProntosanⓇ compress for 15 minutes, subsequent irrigation with distilled water, application of peri-ulcer barrier cream or spray, and the application of ActicoatⓇ on the wound bed. More or less alginate will be applied depending on the amount of exudate. A tertiary dressing of polyurethane foam or bandage will be applied according to the area and the nurse's discretion.
  Other Names: 0,1 % Undecilenamidopropil betaine, 0,1 % Polyhexanide
  Arms: Control group

SUMMARY:
The objective of this clinical trial is to assess the effectiveness of acetic acid in patients suffering from chronic cutaneous ulcers with biofilm. The primary question it seeks to address is whether acetic acid (as a 2% topical solution) is superior to the current standard treatment for chronic cutaneous ulcers with biofilm at our center (Prontosan®).

Participants will be randomly assigned to receive either the acetic acid solution treatment or the standard current treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Continued care (hospital or outpatient) in one of the Consorci Sanitari Alt Penedes i Garraf (CSAPG) units.
* Presence of a cutaneous ulcer with biofilm, with an area of less than 120 cm2, and in any location (except the facial region).
* Plan to undergo treatment and follow-up of the lesion (at least 8 weeks) at the study center.
* Ability to cooperate in necessary evaluations.
* Informed consent for inclusion in the study, either from the participant themselves or from their legal representative.

Exclusion Criteria:

* Participants diagnosed with any of the following conditions:

  1. Ulcers with exposed bone tissue.
  2. Neoplastic-origin ulcers.
  3. Ulcers lasting more than 18 months.
* Participation in another clinical trial involving an experimental intervention during the period of the current trial and/or establishing a visit frequency incompatible with the current trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-04-27 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in ulcer area compared to baseline (percentage) at 8 weeks of treatment | 8 weeks
  The assessment of the ulcer will include measuring its area through digital planimetry.

SECONDARY OUTCOMES:
Percentage of participants with ulcer healing at 4 weeks from the start of treatment. | 4 weeks
  The assessment of the ulcer will performed by the nurse responsible for monitoring the ulcer. The ulcer will be considered fully healed when the surface is epithelialized.
Percentage of participants with ulcer healing at 12 weeks from the start of treatment. | 12 weeks
  The assessment of the ulcer will performed by the nurse responsible for monitoring the ulcer. The ulcer will be considered fully healed when the surface is epithelialized.
Time (days) to ulcer healing from the start of treatment. | up to 12 weeks
  The lesion will be considered fully healed when the surface is epithelialized. This will be confirmed by the nurse responsible for monitoring the lesion.
Changes in the wound bed at 8 weeks according to score of section 6 of the RESVECH2.0 ("Expected Results of the Assessment and Evaluation of Healing of Chronic Wounds" scale. | 8 weeks
  The evaluation of changes will be conducted by a trained nurse to apply the RESVECH 2.0 scale. The scores in Section 6 of the RESVECH scale range from 0 to 14. The higher the score, the greater the severity of the injury.
Number of adverse reactions associated with the treatment, collected from the medical record. | 12 weeks
  The number of adverse reactions will be evaluated through the review of the participant's medical records by a trained member of the research team.
The healthcare expenditure associated with each branch of the study | 12 weeks
  A descriptive analysis of healthcare expenditure associated with each study branch will be conducted using billing data from the center, which is linked to the insured individual's resource utilization.
Change in ulcer area compared to baseline (percentage) at 4 weeks of treatment | 4 weeks
  The assessment of the ulcer will include measuring its area through digital planimetry.
Change in ulcer area compared to baseline (percentage) at 12 weeks of treatment | 12 weeks
  The assessment of the ulcer will include measuring its area through digital planimetry.

CONTACTS AND LOCATIONS:
Overall Officials: Marta De Vicente, Principal Investigator — CSAPG
Locations (1):
- Consorci Sanitari Alt'Pènedes i Garraf, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD (without personal identification data) could be shared by requirement from other researchers after the end of the study, and only for research proposels and previous approval of promotor center of the study (CSAPG). Anyway, Spanish and European Union legal policy about data protection will strictly be followed (IPD will not be transferred outside European Union).
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After publication of main results of the study.
Access Criteria: IPD will be shared only for scientific research purposes and following the Spanish and European Union normative law about data protection. The requirements will be directed to the IP of the study. The IP will evaluate the request to verify and evaluate the data that is requested and the purposes for which it is requested. Next, the IP will transfer the request to the promotor center the study for the final decision.